CLINICAL TRIAL: NCT04043715
Title: Spinal Stimulation for Standing & Walking; Comparison of Transcutaneous & Epidural Stimulation
Brief Title: Comparison of Transcutaneous and Epidural Spinal Stimulation for Improving Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding. PI left the institution
Sponsor: University of Washington (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chet Moritz, Professor, Department of Electrical & Computer Engineering, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004478; EEC-1028725 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Trauma, Nervous System; Wounds and Injuries
Keywords: transcutaneous spinal stimulation; epidural spinal stimulation; physical therapy; lower extremity
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Trauma, Nervous System; Wounds and Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study will compare the benefits of transcutaneous and epidural stimulation in individuals with SCI through a phased intervention program including: 1) baseline testing, 2) PT only, 3) PT + TransQ stimulation, 4) wash out/recovery, 5) PT + Epidural stimulation, 6) follow-up testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Comparison of transcutaneous & epidural stimulation (Other): Comparison of transcutaneous vs epidural electrical stimulation
  Interventions: Device: Transcutaneous spinal stimulation; Device: Epidural spinal stimulation

INTERVENTIONS:
Device: Transcutaneous spinal stimulation — Physical therapy to improve standing and walking
  Other Names: Physical Therapy
Device: Epidural spinal stimulation — Physical therapy to improve standing and walking
  Other Names: Physical Therapy

SUMMARY:
Incomplete spinal cord injuries (SCI) are the most frequent neurologic category, comprising 66.7% of all SCI cases. People with incomplete SCI may retain some ability to move the legs and therefore the capacity to regain walking. Studies that show functional improvement in locomotion via electrical stimulation of lumbosacral circuits suggest that the underlying mechanisms are neuromodulation of lumbosacral spinal cord automaticity and sensory feedback.

Both epidural and transcutaneous spinal stimulation are demonstrating exciting potential to improve limb function for people after chronic SCI. Available treatment options for SCI are less than satisfactory and most often do not achieve full restoration of function. Recent experimental results suggest an exciting new approach of using electrical spinal stimulation to enable users to regain control of their weak or paralyzed muscles. Using surgically-implanted electrodes, epidural stimulation results in remarkable improvements of lower extremity function as well as autonomic functions such as bladder function and sexual function.

In addition to epidural stimulation, over only the last few years a novel strategy of skin surface electrical spinal stimulation has also demonstrated exciting potential for improving walking function. Using a high-frequency stimulation pulse, current can pass through the skin without discomfort and activate the spinal cord; this results in patterned stepping movements for people without SCI and improved lower extremity function following SCI. This study will directly compare skin-surface transcutaneous stimulation with implanted epidural stimulation for improving lower extremity function.

DETAILED DESCRIPTION:
The purpose of this study is to determine the optimal method for delivering spinal stimulation to improve walking in people with incomplete spinal cord injury. By directly comparing non-invasive transcutaneous (TransQ) stimulation with implanted epidural stimulation, investigators hope to guide the field toward the most beneficial method for restoration of lower extremity function. In addition, the investigators may identify subgroups of people that respond better to each type of stimulation, informing personalized treatment for people with different types of spinal cord injury. The research team will explore the following specific aims:

Aim 1: Evaluate the improvements in lower extremity and autonomic function via transcutaneous spinal stimulation and intensive physical therapy for people with chronic SCI.

Aim 2: Quantify additional improvements in lower extremity and autonomic function via epidural spinal stimulation and intensive physical therapy for people with chronic SCI.

The investigators will test the hypothesis that epidural stimulation leads to greater improvements than an equal dose of transcutaneous stimulation. To compare these 2 stimulation methods the study team will evaluate voluntary control of muscle activity via EMG and kinematic parameters of locomotion, as well as improvements in bladder and other autonomic functions and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. have a spinal cord injury at least one-year duration;
2. are between 21 and 70 years of age;
3. have difficulty with leg functions and mobility in activities of daily living (e.g. walking, transferring surface to surface, standing);
4. are candidates for an implanted stimulator;
5. are willing and able to have surgical implantation of the epidural stimulator for the treatment of pain according to the study timeline;
6. experience chronic pain;
7. are in stable medical condition without cardiopulmonary disease or frequent autonomic dysreflexia that would contraindicate participation in lower extremity rehabilitation or testing activities;
8. are capable of performing simple cued motor tasks;
9. have the ability to attend 3-5 sessions per week physical therapy sessions and testing activities over three months;
10. have adequate social support to be able to participate in assessment sessions occurring between once per week to once per month for up to 9 months;
11. are volunteering to be involved in this study;
12. are cleared for gait training by primary physician of the subject;
13. and have ability to read and speak English

Exclusion Criteria:

1. have autoimmune etiology of spinal cord dysfunction/injury;
2. have a history of additional neurologic disease, such as stroke, MS, traumatic brain injury, etc.;
3. have peripheral neuropathy (diabetic polyneuropathy, entrapment neuropathy, etc.);
4. have rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.);
5. have significant medical disease; including uncontrolled systemic hypertension with values above 170/100 mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation;
6. have active cancer;
7. have cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention;
8. have unhealed fracture, contracture, pressure sore, or urinary tract infection or other illnesses that might interfere with lower extremity rehabilitation or testing activities;
9. have any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician;
10. are pregnant;
11. are dependent on ventilation support;
12. have implanted stimulator (e.g. epidural stimulator, vagus nerve stimulator, pacemaker, cochlear implant, etc.);
13. have depression or anxiety based on the Center for Epidemiologic Studies Depression Scale (CESD) (score >16/60) and General Anxiety Disorder-7 item Questionnaire (score >9/21), respectively.
14. have alcohol and/or drug abuse;
15. have cognitive impairment based on Short Portable Mental Status Questionnaire (SPMSQ) (score >2/10);
16. are unable to read and/or comprehend the consent form;
17. are unable to understand the instructions given as part of the study;
18. have established osteoporosis and are taking medication for osteoporosis treatment;
19. have bone mineral density T scores ≤ -2.0 in anteroposterior lumbar spine and/or proximal femur measured by DEXA (if participants are clear for other criteria and have not been examined by DEXA at the screening, we will ask participants to undergo DEXA to reveal any risk of weight bearing activity);
20. have a low-energy fracture history before or after spinal cord injury;
21. have a history of orthopedic surgery in lower extremities that may be a confounding factor for interpretation of the results (such as tendon transfer, tendon or muscle lengthening for spasticity management, etc.);
22. have fixed lower extremity joint contractures;
23. are taller than 80 inches and/or weighs more than 350 pounds (due to the limitation of the experimental equipment such as the body weight support system);
24. lack the ability to fully comprehend and/or perform study procedures in the investigator's opinion/judgement

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Neuromuscular Recovery Scale | 8-11 months
  Neuromuscular recovery scale is an assessment for sitting, standing and walking functions based on a comparison to pre-injury performance criteria or how a task was performed one day prior to spinal cord injury and without use of compensation strategies. The items consists of stand retraining, stand adaptability, step retraining, step adaptability, sit, reverse sit up, trunk extension in sitting, sit to stand , stand, walking, and upper limb functions. They are score the scale of 4 based on how close to the function in the pre-injured condition.

SECONDARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Examination | 8-11 months
  Standard neurologic examination that is routinely used to determine the levels and severity of spinal cord injury. Includes manual muscle strength testing and dermatomal light touch and pin prick sensory examination.
Somatosensory evoked potentials | 8-11 months
  Measurement of amplitude of electrical potentials that is recorded by surface electrodes over the scalp following electrical stimulation of peripheral nerve from the wrist. The amplitude of the response is reported in micro-volts.
Motor evoked potentials - Latency | 8-11 months
  Measurement of latency of electrical potentials that is recorded by surface electrodes over the skin of limb muscles following spinal stimulation or magnetic stimulation of brain over the scalp. The latency of the response is reported in micro-seconds.
Motor evoked potentials - Amplitude | 8-11 months
  Measurement of amplitude of electrical potentials that is recorded by surface electrodes over the skin of limb muscles following spinal stimulation or magnetic stimulation of brain over the scalp. The amplitude of the response is reported in micro-volts.
Berg Balance Test | 8-11 months
  Measurement of balance in standing and sitting. The balance score consists of 14 items and is reported in the scale of 56 (each items are score in 0-4).
Six-minute walk test | 8-11 months
  Measurement of walking ability. The distance is reported in meter.
Ten-minute walk test | 8-11 months
  Measurement of walking ability. The walking speed is reported in meter per second.
Kinetic and kinematic gait analysis using 3D camera system - angle | 8-11 months
  Measurement of leg function and walking ability. Joint angle is reported in degree angle.
Kinetic and kinematic gait analysis using 3D camera system - velocity | 8-11 months
  Measurement of leg function and walking ability. Velocity is reported in meter per second.
Electromyography recording of LE and trunk muscles | 8-11 months
  Measurement of muscle and nerve functions. The muscle activities are reported in micro-volts.
Spinal Cord Injury - Quality of Life (SCI-QOL) questionnaire | 8-11 months
  Patient reported quality of life scale. The SCI-QOL consists of 19 item banks, and is reported by T-score comparing the mean of the functional level in the population.
Spinal Cord Injury - Functional Index (SCI-FI) questionnaire | 8-11 months
  Patient reported functional scale. The SCI-QOL consists of 10 item banks, and is reported by T-score comparing the mean of the functional level in the population.
Wartenberg Pendulum Test | 8-11 months
  The Wartenberg Pendulum Test is a measure of spastic hypertonia. Using computer data for number of oscillations and amplitude, values of the Relaxation index (R1 and R2) are calculated and compared to norms.
Walking Index for Spinal Cord Injury II | 8-11 months
  A functional capacity scale designed to measure improvements in ambulation in persons with spinal cord injury, by evaluating the amount of physical assistance, braces or devices required to walk 10 meters.
Neurogenic Bladder Symptom Score | 8-11 months
  24-item questionnaire designed to assess bladder symptoms in patients with neurogenic bladder dysfunction as a result of spinal cord injury, multiple sclerosis, and spinal bifida.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Saigal, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States